CLINICAL TRIAL: NCT02157961
Title: Doc's Health - Doctor as a Patient - An Observational Study on Health Behavior of Physicians in Germany
Brief Title: Doctor's Health - Health Behavior of Physicians in Germany
Acronym: Doc'sHealth
Status: Completed | Type: Observational
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Jochen Gensichen, MD, MA, MPH, professor, University of Jena
Other Study IDs: 4058-04/14
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Diseases; Chronic Illnesses
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- General Practitioner / Family Physician in German Primary care
- Medical Specialists: Working in the ambulatory setting

SUMMARY:
This is an observational study to assess the health behavior of Physicians from medical practices in Germany. Physicians will be asked by a questionnaire (self-report) on health behavior, self-diagnostics and self-medication in case of sickness. We will send the questionnaire to 1000 General Practitioners and to 300 medical specialists in Germany. We expect a response rate of 25-30 %. After electronically data-entry we will run a descriptive analysis for primary outcome. Results may provide a better understanding of the Physicians health behavior.

ELIGIBILITY:
Inclusion Criteria:

* Physicians in German ambulatory setting

Exclusion Criteria:

* any

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physicians in Germany
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2014-04; Primary Completion 2014-11 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Physicians health behavior | 1 day
  questionnaire

SECONDARY OUTCOMES:
Physicians medication use | 1 day
  questionnaire
Physicians preventive care | 1 day
  questionnaire

OTHER OUTCOMES:
Locus of internal control | 1 day
  questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of General Practice, University of Jena, Jena, Germany

REFERENCES:
- See also: Click here for more information about this study — http://www.allgemeinmedizin.uni-jena.de